CLINICAL TRIAL: NCT00761007
Title: Double-blind, Randomised, Placebo-controlled, Parallel Group Study to Evaluate the Effect of a 4-week Treatment With Oral Doses of Ibodutant (Code: MEN15596) in Irritable Bowel Syndrome (IBS).
Brief Title: Ibodutant for Relief of Irritable Bowel Syndrome (IRIS)
Acronym: IRIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NAK 03; 2008-000214-71 (EudraCT Number)
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Bowel disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Intestinal Diseases | interventions — ibodutant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ibodutant 10 mg (Experimental)
  Interventions: Drug: Ibodutant
- Ibodutant 30 mg (Experimental)
  Interventions: Drug: Ibodutant
- Ibodutant 60 mg (Experimental)
  Interventions: Drug: Ibodutant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibodutant — Oral tablet, dose level 1 (10 mg), once daily
  Other Names: Code: MEN 15596
  Arms: Ibodutant 10 mg
Drug: Ibodutant — Oral tablet, dose level 2 (30 mg), once daily
  Other Names: Code: MEN 15596
  Arms: Ibodutant 30 mg
Drug: Ibodutant — Oral tablet, dose level 3 (60 mg), once daily
  Other Names: Code: MEN 15596
  Arms: Ibodutant 60 mg
Drug: Placebo — Oral tablet matching the three dose levels of ibodutant, once daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the benefit of treatment with oral dose of Ibodutant (code: MEN 15596) on IBS symptoms and the safety and tolerability of this therapy.

DETAILED DESCRIPTION:
Irritable Bowel Syndrome (IBS) is a functional disorder characterised by chronic or recurrent abdominal pain or discomfort associated with altered bowel habits. This trial aims to evaluate the efficacy of Ibodutant in improvement of IBS symptoms through a daily oral administration, testing three dosages or placebo in IBS patients for 4-weeks. In each patient, the experimental clinical phase encompasses a screening/ 2-week run-in period (no study medication), followed by a 4-weeks treatment period and a 2-weeks treatment withdrawal period, for total study duration of 8 weeks in each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 - 70 years.
2. Clinical diagnosis of IBS .
3. For patients older than 50 years or patients with positive family history of colorectal cancer: normal results from colonoscopy or flexible sigmoidoscopy.
4. Use of appropriate contraceptive methods.
5. Normal physical examination or without clinically relevant abnormalities.

Exclusion Criteria:

1. Patients with organic abnormalities of the gastro-intestinal tract including history of colonic or major abdominal surgery, current or previous diagnosis of neoplasia, inflammatory bowel diseases, symptomatic gallbladder stone disease, diverticulosis/diverticulitis, ectopic endometriosis.
2. History of gluten enteropathy.
3. Lactose intolerance as assessed by response to diet
4. Diagnosis of ova or parasites, or occult blood in the stool in the previous 6 months.
5. Previous diagnosis of Diabetes Mellitus (either type 1 or 2)
6. Unstable medical condition.
7. Concomitant medication within 7 days prior to screening with drugs known to interfere with gastro-intestinal motility and sensitivity.
8. Pregnancy or breastfeeding.
9. Patient not able to understand or collaborate throughout the study.
10. Participation in other clinical trials in the previous 4 weeks.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2008-07; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Study Chair — Department of Gastroenterology, University Hospital Katholieke Universiteit Leuven, Belgium
Locations (6):
- Center for Clinical and Basic Research (CCBR), Ballerup Municipality, Denmark
- emovis GmbH, Berlin, Germany
- Digestive Diseases Center "Gastro", Riga, Latvia
- Federal State Institution "Outpatient clinic #3" of President's Management Department of the Russian Federation, Moscow, Russia
- Academy of Medical Science of Ukraine, Dnipropetrovsk, Ukraine
- Synexus Midlands Clinical Research Centre, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 15/07/2008, last subject observed 18/02/2009, at 60 study centres in 9 European countries (Denmark, Germany, Italy, Latvia, Russia, Slovak Republic, Spain, United Kingdom, and Ukraine.
Pre-assignment Details: Subjects underwent a 2-week screening period to meet inclusion/exclusion criteria and were subsequently randomised.
Groups:
- Ibodutant 10 mg; Ibodutant 30 mg; Ibodutant 60 mg; Placebo: oral tablet, once daily
Period: Overall Study
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Started | 142 | 135 | 139 | 138
Safety (>=1 Dose of Study Medication) | 140 | 135 | 139 | 137
ITT (>= 1 Assessment Post-Randomisation) | 140 | 133 | 135 | 136
Completed | 129 | 124 | 121 | 131
Not Completed | 13 | 11 | 18 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo | Total
Number analyzed (Participants) | 140 | 133 | 135 | 136 | 544
Age Continuous [Mean (Standard Deviation); unit: years] | 43.9 (13.43) | 45.0 (12.66) | 44.4 (12.97) | 43.7 (13.73) | 44.2 (13.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 79 | 90 | 94 | 367
  Male | 36 | 54 | 45 | 42 | 177
IBS-Subtype [Number; unit: participants]
  IBS-Diarrhea | 68 | 53 | 59 | 54 | 234
  IBS-Constipation | 37 | 44 | 34 | 50 | 165
  IBS-Mixed | 26 | 29 | 34 | 22 | 111
  IBS-Unsubtyped | 9 | 7 | 8 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Response of Overall IBS Symptom Relief - 50% Rule
Description: Weekly binary question (yes/no): "Did you have satisfactory relief of your overall IBS symptoms since the last visit?"
  Responder: report of satisfactory overall IBS symptom relief = "Yes" 2/4 weeks (50% rule)
Time Frame: Four weeks
Population: Intention-to-Treat (N=544)
Measure: Number; unit: Participants
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Number analyzed (Participants) | 140 | 133 | 135 | 136
Participants | 79 | 61 | 61 | 78

2. Secondary Outcome: Response of Overall IBS Symptom Relief - 75% Rule
Description: Weekly binary question (yes/no): "Did you have satisfactory relief of your overall IBS symptoms since the last visit?"
  Responder: report of satisfactory overall IBS symptom relief = "Yes" 3/4 weeks (75% rule)
Time Frame: Four weeks
Population: Intention-to-Treat (N=544)
Measure: Number; unit: Participants
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Number analyzed (Participants) | 140 | 133 | 135 | 136
Participants | 53 | 39 | 37 | 48

3. Post Hoc Outcome: Response of Overall IBS Symptom Relief in the Subgroup of Patients With IBS-Diarrhea (IBS-D) and Pain at Baseline - 75% Rule
Description: as for outcome 2
Time Frame: Four weeks
Population: Intention-to-treat subgroup of patients with IBS-D and baseline pain score>1 (in a 5-point scale ranging from 0=no pain to 4=very severe) (N=189)
Measure: Number; unit: Participants
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Number analyzed (Participants) | 54 | 43 | 48 | 44
Participants | 31 | 15 | 17 | 19

4. Secondary Outcome: Response of Overall IBS Symptom Relief in the Subgroup of Patients With IBS With Diarrhea (IBS-D) - 75% Rule
Description: as for outcome 2
Time Frame: Four weeks
Population: Intention-to-treat (ITT) subgroup of patients with IBS-D (N=234)
Measure: Number; unit: Participants
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Number analyzed (Participants) | 68 | 53 | 59 | 54
Participants | 33 | 17 | 22 | 25

ADVERSE EVENTS:
Time Frame: Four weeks
Description: Analysed for the Safety Population (all patients who took at least one dose of study medication, N=551)
Arm/Group | Ibodutant 10 mg | Ibodutant 30 mg | Ibodutant 60 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/140 | 3/135 | 1/139 | 0/137
Other Adverse Events (participants affected / at risk) | 29/140 | 29/135 | 28/139 | 26/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg (N=140) | Ibodutant 30 mg (N=135) | Ibodutant 60 mg (N=139) | Placebo (N=137)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibodutant 10 mg (N=140) | Ibodutant 30 mg (N=135) | Ibodutant 60 mg (N=139) | Placebo (N=137)
Abdominal pain (Gastrointestinal disorders) | 4 (5) | 5 (5) | 5 (5) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 1 (1) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (12) | 3 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 9 (12) | 7 (10) | 5 (6) | 8 (10)
Nasopharyngitis (Infections and infestations) | 5 (6) | 6 (7) | 4 (4) | 7 (9)
Nausea (Gastrointestinal disorders) | 5 (5) | 6 (7) | 3 (3) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less